CLINICAL TRIAL: NCT06675253
Title: Perioperative Fluid Therapy from the Perspective of an Anesthesiologist
Acronym: PFT
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Other Study IDs: Fluid_Therapy_MP
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2022-04

CONDITIONS: Perioperative Care
Keywords: Fluid therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A survey conducted in 2022 in ,,Medycyna Praktyczna'' magazine, publishing house regarding fluid therapy in hospital wards showed that many recommendations regarding proper fluid therapy have become common practice, but there are still a significant number of practices established over the years that differ significantly from the principles of good clinical practice

DETAILED DESCRIPTION:
In the period August 28, 2021- April 15, 2022, two online surveys were conducted among anesthesiologists in the ,,Practical Medicine'' magazine, asking about the principles they follow when conducting PFT(Perioperative Fluid Therapy).

ELIGIBILITY:
Inclusion Criteria:

* medical physician

Exclusion Criteria:

* no medical physician

Min Age: 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: survey study conducted among doctors
Sampling Method: Non-Probability Sample
Enrollment: 913 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
evaluation of clinical practice | 8 months from the publication of the survey
  survey results showing how clinicians conduct fluid therapy in the perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No